CLINICAL TRIAL: NCT04500990
Title: Magnetic Resonance Imaging (MRI) Diffusion-weighted Imaging (Dwi) None-Gaussian Model Predicting Early Response to Immunotherapy in Digestive System Malignancies: a Prospective Observational Study
Brief Title: MRI DWI None-Gaussian Model Predicting Early Response to Immunotherapy in Digestive System Malignancies: a Prospective Observational Study
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Peking University (Other)
Responsible Party: Principal Investigator, Shen Lin, professor, Peking University
Other Study IDs: MRI immunotherapy
Record Dates: First submitted 2020-07-30; First posted 2020-08-06 (Actual); Last update posted 2020-08-06 (Actual); Status verified 2020-07

CONDITIONS: Immunotherapy; Digestive System Neoplasm
Keywords: MRI; DWI; Digestive system malignancies; Early response
MeSH Terms: conditions — Digestive System Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Single agent PD-1/PD-L1 inhibitor: Patients will receive single agent PD-1/PD-L1 inhibitor in a predefined group.
  Interventions: Radiation: MRI test
- Combined immunotherapy: Patients will receive combined immunotherapy in a predefined group. PD-1/PD-L1 inhibitor will be combined with target therapy, such as lenvatinib, enrotinib, herceptin et al.
  Interventions: Radiation: MRI test

INTERVENTIONS:
Radiation: MRI test — Patients will receive diagnostic MRI test on d0.
Radiation: MRI test — Patients will receive diagnostic MRI test on d8±1.
Radiation: MRI test — Patients will receive diagnostic MRI test on d30±2.

SUMMARY:
This is a prospective two cohorts observational study aimed to investigate the predicting value of MRI none-Gaussian model in digestive malignancies patients who received single agent PD-1/PD-L1 inhibitor or combined immunotherapy.

ELIGIBILITY:
Inclusion Criteria:

* age ≥ 18 years, ECOG 0-1, expected survival ≥3 months;
* pathologically confirmed digestive system adenocarcinoma, including but not restricted to gastric adenocarcinoma, colorectal cancer, pancreatic adenocarcinoma et al;
* pathologically confirmed PD-L1 expression, or MMR-deficient (dMMR)/microsatellite instability (MSI-H) or high tumor mutation burden (TMB-H) or other indication for immunotherapy;
* at least one target lesion, if there is no target lesion the thickness of cavity viscera lesion should exceed 1cm;
* patients will receive single agent PD-1/PD-L1 inhibitor, or combined immunotherapy such as: lenvatinib, enrotinib or herceptin;
* screening laboratory values must meet the following criteria: hemoglobin ≥ 9.0 g/dL; neutrophils ≥ 1500 cells/ μL; platelets ≥ 100 x 10^3/ μL; total bilirubin ≤ 2.0 x upper limit of normal (ULN); aspartic transaminase (AST) and alanine transaminase (ALT) ≤ 2.5 x ULN without, and ≤ 5 x ULN with hepatic metastasis; serum creatinine ≤1.5 x ULN, and serum creatinine rate >50μmol/L; activated partial thromboplastin time (APTT)、international normalized ratio (INR), prothrombin lime (PT)≤1.5×ULN;
* echocardiography: left ventricular ejection fraction≥50%
* volunteer participate, signed written informed consent form.

Exclusion Criteria:

* claustrophobia or other contraindication for MRI testing;
* received prior anti-PD-1/PD-L1 or other immune checkpoint inhibitors;
* combined immunotherapy contains chemotherapy agent;
* contain other histology component except adenocarcinoma；
* hypersensitivity after other monoclonal antibody infusion；
* coexist other malignancy in last five years;
* active autoimmune disease, or who received systemic treatment with corticosteroids (> 10 mg daily prednisone equivalent) or other immunosuppressive medications within 2 weeks of first dose;
* Cavity effusion (pleural effusion, ascites, pericardial effusion, etc.) are not well controlled, and need locally treatment or repeated drainage;
* obvious bleeding tendency or had CTCAE≥3 grade；
* subjects are eligible with clinically controlled and stable neurologic function ≥ 4 weeks, which is no evidence of CNS disease progression; subjects with spinal cord compression and cancerous meningitis are not eligible；
* vaccination within 28 days of the first administration of trial treatment.

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Patients receive treatment in Beijing Cancer Hospital.
Sampling Method: Non-Probability Sample
Enrollment: 40 (Estimated)
Dates: Start 2020-09 (Estimated); Primary Completion 2021-07 (Estimated); Study Completion 2021-07 (Estimated)

PRIMARY OUTCOMES:
Objective Response Rate | from enrollment of the first subject until the database cut-off approximately 12 months later.
  The rate of patients reached complete response or partial response.

SECONDARY OUTCOMES:
Progress free survival | from enrollment of the first subject until the database cut-off approximately 12 months later.
  the time from enrollment to disease progression or death or loss of follow-up.
Overall survival | from enrollment of the first subject until the database cut-off approximately 12 months later.
  the time from enrollment to death or loss of follow-up.

CONTACTS AND LOCATIONS:
Overall Officials: Lin Shen, professor, Principal Investigator — Peking University
Locations (1):
- Beijing Cancer Hospital, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: No